CLINICAL TRIAL: NCT06420505
Title: Multicenter Observatory Evaluating the Polymer-Free Sirolimus Eluting Coronary Stent System VIVO ISAR in Routine Clinical Practice (CELEBRITY Observatory)
Brief Title: Evaluation of the Vivo Isar Stent System in Routine Clinical Practice
Acronym: CELEBRITY
Status: Recruiting | Type: Observational
Sponsor: Translumina GmbH (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: TRANSLUMINA
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Artery Coronary Stenosis
MeSH Terms: conditions — Coronary Stenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — The Vivo ISAR is indicated for improving coronary luminal diameter in patients with symptomatic ischemic heart disease.

SUMMARY:
The rationale for this observatory is to evaluate clinical outcomes and collect data of the Polymer Free Sirolimus Eluting Coronary Stent System in Real World CAD Patients with follow-up at 12 months. All medications and procedures to be used/ performed in this observatory are commonly used/performed for clinical indications as part of standard of care and have well-defined safety profiles.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Ability to provide signed informed consent form.
* Male or non-pregnant female patient (Pregnancy status to be confirmed verbally from the female patient of reproductive age)
* Presentation with acute coronary syndrome or chronic coronary syndrome with stable angina or angina equivalent symptoms or with a positive noninvasive test for ischemia or evidence of a functionally significant coronary stenosis.
* Patient having social security number.
* Patient treated only with Vivo ISAR stent in case of single or multiple vessel stenting

Exclusion Criteria:

* Concurrent participation in another clinical trial.
* Having benefited from an angioplasty of ≤ 1 month with a stent other than Vivo ISAR.
* Planned elective surgery in next 6 months
* Cardiogenic shock/ hemodynamically unstable patients
* Concurrent medical condition with a life expectancy of less than 12 months
* History of cerebrovascular accident in the last 6 months.
* Vulnerable patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all-comers population who qualify for percutaneous coronary intervention (consisting of patients with symptomatic coronary artery disease including chronic coronary syndromes (CCS) and ACS) of any gender, ≥ 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-11-29 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
rate of target lesion failure | 12 months post-procedure
  • The rate of target lesion failure at 12 months follow-up defined as the composite endpoint of:
  * Cardiac death
  * Myocardial infarction related to the target vessel
  * Clinically documented target lesion revascularization

SECONDARY OUTCOMES:
Device success rate | 12 months post-procedure
  • Device success rate defined as successful placement and deployment of the device at the target lesion site with successful removal of the delivery system leaving a final residual stenosis <30% of the segment of the culprit lesion covered by the stent at 1 year
Procedural success rate | 7 days post-procedure
  * Procedural success rate defined as device success without major ischemia-related adverse cardiac events during hospitalization and up to a maximum of 7 days post-procedure :
  * Cardiac death
  * Any MI
  * Target-vessel MI
Assess reperfusion | 12 months post-procedure
  Target Lesion Revascularization at 12 months
• Evaluate the antiplatelet treatment | 12 months post-procedure
  antiplatelet consumption during 1 year after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Thibault Lhermusier, Pr, Principal Investigator — University Hospital, Toulouse
Locations (19):
- France (19):
  - Clinique Axium, Aix-en-Provence
  - CHU CAEN, Caen
  - Hôpital A. Schweitzer - GHCA, Colmar
  - Clinique Louis Pasteur, Essey-lès-Nancy
  - CH Haguenau, Haguenau
  - CHU La Timone, Marseille
  - Hopital Nord, Marseille
  - HP Jacques Cartier, Massy
  - Clinique Pont de Chaume, Montauban
  - Hôpital Privé du Confluent, Nantes
  - Polyclinique Les Fleurs, Ollioules
  - APHP, Paris
  - HP Claude Galien, Quincy-sous-Sénart
  - CHU Reims, Reims
  - Clinique Saint Hilaire, Rouen
  - CHRU Strasbourg, Strasbourg
  - CH de Bigorre, Tarbes
  - Clinique Pasteur, Toulouse
  - Chu Toulouse, Toulouse